CLINICAL TRIAL: NCT03290027
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled Study of the Safety and Efficacy of DFD-03 Lotion in the Treatment of Acne Vulgaris for 12 Weeks
Brief Title: A Study of the Safety and Efficacy of DFD-03 for the Treatment of Acne Vulgaris
Acronym: DFD-03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFD-03-CD-005
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Results first posted 2020-05-26 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): DFD-03 (0.1% tazarotene) Lotion
  Interventions: Drug: DFD-03
- Vehicle (Placebo Comparator): Vehicle (0% tazarotene) Lotion
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: DFD-03 — DFD-03 Lotion
  Other Names: Tazarotene 0.1% Lotion
  Arms: Active
Other: Placebo Comparator — Vehicle (tazarotene 0%) Lotion
  Other Names: Vehicle
  Arms: Vehicle

SUMMARY:
Enrollment of subjects with mild to moderate facial acne. Efficacy was assessed by using an Investigator's Global Assessment scale (IGA 5 point scale) and by counting the number of inflammatory and non-inflammatory lesions on the face at Baseline and Weeks 4, 8, and 12.

Safety assessments included the investigator's assessment of local cutaneous tolerance of the treated skin (dryness, non-lesional erythema, peeling, stinging, burning, and itching, vital signs, and adverse events (AEs).

DETAILED DESCRIPTION:
Enrollment of subjects with mild to moderate facial acne. Subjects with acne lesions of any severity on the chest and/or back (including shoulders) were enrolled provided they had mild to moderate acne on the face. During the 12-week treatment period subjects used the study product twice daily. Subjects were instructed to treat the entire face (and chest and/or back including shoulders, if applicable).

Efficacy was assessed by using an Investigator's Global Assessment scale (IGA 5 point scale) and by counting the number of inflammatory and non-inflammatory lesions on the face at Baseline and Weeks 4, 8, and 12.

Safety assessments included the investigator's assessment of local cutaneous tolerance of the treated skin (dryness, non-lesional erythema, peeling, stinging, burning, and itching; assessed separately on the chest and/or back including shoulders (if applicable), vital signs (blood pressure and pulse rate), and adverse events (AEs). Urine pregnancy tests were performed at Baseline and at every visit through Week 12 for all female subjects. A physical examination was performed.

ELIGIBILITY:
Main Inclusion Criteria:

1. Subject must be at least 9 years of age.
2. A clinical diagnosis of mild to moderate facial acne vulgaris.
3. Inflammatory lesion count (papules and pustules) of at least 20 on the face, Non-inflammatory lesion count (closed and open comedones) of at least 25 on the face and No more than 2 nodulocystic lesions on the face.
4. Females, regardless of childbearing potential, if sexually active, must be on or use an acceptable method of birth control.
5. Subject must be in good general health as determined by the investigator and supported by medical history, physical and Vital Signs exam.

Main Exclusion Criteria:

1. Females who are pregnant or lactating or planning to become pregnant.
2. Treatment with the following products:

   1. Topical acne treatments or other topical facial medication on the treatment area.
   2. Systemic corticosteroids, systemic acne treatments including systemic antibiotics used for treatment of acne.
   3. Systemic retinoid use.
   4. Undertaken certain facial procedures such as chemical peel, laser treatment, photodynamic therapy, acne surgery, cryodestruction or chemodestruction, x-ray therapy, intralesional steroids, dermabrasion, or depilation (except eyebrow shaping).
   5. Treatment with a medication or procedure that, in the opinion of the investigator, would put the subject at unacceptable risk for participation in the study or may interfere with evaluations in the study.
   6. Treatment with an investigational product or device in the 30 days.
3. Known allergic reaction to retinoids or tazarotene.
4. Presence of any facial skin disease or condition that would interfere with the study or place the subject at unacceptable risk including sunburn, rosacea, seborrheic dermatitis, perioral dermatitis, lupus, dermatomyositis, psoriasis, eczema, squamous cell carcinoma, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, bacterial folliculitis or any other facial disease or condition.
5. Subjects with a serious and/or chronic medical condition such as chronic or active liver disease, renal impairment, heart disease, severe respiratory disease, rheumatoid arthritis, current malignancies, immunocompromised conditions, or any other disease that, in the opinion of the investigator, would interfere with the study or place the subject at unacceptable risk.
6. Subjects who have been in another investigational trial within 30 days.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, M.D., Study Director — Dr. Reddy's Laboratories Inc.
Locations (1):
- Dr. Seemal, Plano, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Vehicle
Started | 277 | 273
Completed | 219 | 228
Not Completed | 58 | 45

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) - The ITT population was the primary efficacy analysis data set and consisted of all subjects who were randomized and dispensed study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Vehicle | Total
Number analyzed (Participants) | 277 | 273 | 550
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 91 | 91 | 182
  Between 18 and 65 years | 186 | 182 | 368
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.2 (7.9) | 21.1 (8.0) | 21.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 158 | 303
  Male | 132 | 115 | 247
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 109 | 105 | 214
  Not Hispanic or Latino | 168 | 168 | 336
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 14 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 58 | 109
  White | 200 | 194 | 394
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 277 | 273 | 550

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in the Inflammatory Lesion Counts on the Face
Description: Change in inflammatory lesion counts on the face from baseline to Week 12 - will be analyzed using a two way analysis of covariance (ANCOVA) model
Time Frame: Baseline to Week 12
Population: Intent To Treat (ITT) Population - All subjects randomized and dispensed study medication.
Measure: Mean (Standard Deviation); unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 277 | 273
Number analyzed (Lesions) | 277 | 273
Lesions
  Baseline | 30.1 (9.81) | 29.8 (9.13)
  Week 12 | 15.4 (11.43) | 16.9 (11.78)

2. Primary Outcome: Absolute Change in the Non-inflammatory Lesion Counts on the Face
Description: Change in non-inflammatory lesion counts on the face from baseline to Week 12 - will be analyzed using the same ANCOVA model
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 277 | 273
Lesions
  Baseline | 37.4 (14.71) | 36.6 (13.07)
  Week 12 | 20.3 (13.88) | 22.1 (18.26)

3. Primary Outcome: Proportion of Subjects With Treatment Success Based on IGA Score
Description: IGA success at Week 12 (an IGA score of 0 (Clear) or 1 (almost clear) with at least a 2-grade reduction from baseline) - will be analyzed using the Cochran-Mantel-Haenszel (CMH) test for general association
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 277 | 273
Participants | 51 | 34

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time treatment was initiated until study product treatment was discontinued, except for spontaneously reported SAEs, which were to be reported up to 30 days after discontinuing study product use.
Arm/Group | Active | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/273
Serious Adverse Events (participants affected / at risk) | 2/277 | 1/273
Other Adverse Events (participants affected / at risk) | 0/277 | 0/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=277) | Vehicle (N=273)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) — Worsening of Anxiety
Polyps/Epithelioid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Overian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT03290027/Prot_SAP_000.pdf